CLINICAL TRIAL: NCT00217893
Title: ETS Reduction in High-Risk Preteens: A Controlled Trial
Brief Title: Environmental Tobacco Smoke Exposure Reduction in High-Risk Preteens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melbourne Hovell, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 293; R01HL066307 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Combination of counseling, cotinine feedback, and contingent incentives.
  Interventions: Behavioral: Counseling; Behavioral: Urine Cotinine Feedback; Behavioral: Contingent Incentives
- 2 (Active Comparator): Usual education program
  Interventions: Behavioral: Usual education program

INTERVENTIONS:
Behavioral: Counseling — One-on-one behavioral counseling with pre-teen child; 8 to 10 weekly or bi-weekly sessions; focus on identifying sources of exposure to ETS and means to avoid exposure; goal-setting, role-playing, monitoring progress, feedback includes reported info and urine cotinine level.
  Arms: 1
Behavioral: Urine Cotinine Feedback — Urine collected from child at each weekly/bi-weekly counseling session; cotinine level discussed at subsequent session.
  Arms: 1
Behavioral: Contingent Incentives — Child earns small prizes for on-task behavior in sessions, plus earns tokens redeemable for other prizes based on reduction in ETS exposure (reported and cotinine level).
  Arms: 1
Behavioral: Usual education program — Participants will receive the usual education about ETS.
  Arms: 2

SUMMARY:
This study will determine the effect of combining counseling, urine cotinine feedback, and incentives in reducing environmental tobacco smoke (ETS) exposure and susceptibility to smoking among high-risk preteens.

DETAILED DESCRIPTION:
BACKGROUND:

Parent counseling reduced children's ETS exposure in previous studies. This study will determine if interventions directed to preteens alone can reduce ETS exposure. The original pilot study showed that counseling reduced preteen's ETS exposure. New analyses showed that counseling reduced exposure to preteens in the NIH asthma study. A third pilot study showed that counseling plus feedback and incentives reduced preteens' ETS exposure. Based on these results, the number of counseling sessions were decreased to 10, inclusion criteria were liberalized, and recruitment sources were added to assure feasibility.

DESIGN NARRATIVE:

This study will determine the effect of combining counseling, feedback, and incentives on reducing second hand smoke (SHS) exposure and susceptibility to smoking among high-risk preteens. Two hundred youth aged 8 to 13 years old, including African American, Latino, Anglo, and other racial/ethnic groups, will be recruited. Preteens must be nonsmokers who are exposed to ETS in their home. Youth will be recruited sequentially and assigned to usual education or a combination of counseling, cotinine feedback, and contingent incentives. Outcome measures will be obtained prior to intervention, and at Months 5, 9, and 12. Preteens in the intervention condition will receive eight in-home counseling sessions and seven phone counseling sessions over a 5-month period. Urine samples will be analyzed for cotinine using highly sensitive (detection limit .05 ng/ml) and reliable procedures as employed by CDC (ID-LC/MS/MS). The same measures will be used for cotinine feedback for preteens in the intervention condition. Repeated measures analyses of differential exposure to ETS will be employed. Mixed effect regression (REML) and generalized estimating equations (GEE) models will be used for outcome analyses. Exploratory analyses will address questions about the environmental and social determinants of tobacco use and ETS exposure based on the researcher's Behavioral Ecological Model.

Primary objectives include the following: 1) to determine whether counseling plus cotinine feedback and incentives reduces ETS exposure more than does usual tobacco control education (measured by self-report ETS exposure by preteen and parent, and preteen urine cotinine at Month 5); and 2) to determine whether the experimental condition results in differential maintenance in ETS exposure-reduction compared to usual tobacco control education during follow-up (measured by self-report ETS exposure by preteen and parent, and preteen urine cotinine at Months 9 and 12).

Secondary objectives include the following: 1) to explore whether there is a differential rate of cigarette experimentation between groups; to explore whether there is a differential rate of experimentation with alcohol/drugs among groups; 2) to explore the differential level of tobacco use "susceptibility" among experimental groups; 3) to explore the degree to which youth avoid ETS exposure from family members and friends; and 4) to explore the multiple social and possible genetic factors that are independent and in combined association with ETS exposure and change in exposure (measured by preteen and parent self-report at Months 5, 9, and 12).

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking preteen
* Resides in San Diego county
* Smoker lives in the household
* Exposed to an average of 2 cigarettes per day over the week prior to study entry OR urine cotinine greater than or equal to 2.0 ng/mL

Exclusion Criteria:

* Preteen who has smoked in the 30 days prior to study entry or who has smoked more than 10 cigarettes within lifetime

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2003-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
ETS exposure | Measured from baseline to 5 months
Maintenance in ETS exposure-reduction | Measured 5, 9, and 12 months post-baseline

SECONDARY OUTCOMES:
Tobacco use experimentation | Measured from baseline through 5, 9, and 12 months
Experimentation with alcohol/drugs | Measured from baseline through 5, 9, and 12 months
Avoidance of ETS exposure from family members and friends | Measured from baseline through 5, 9, and 12 months
Multiple social and possible genetic factors that are independent and in combined association with ETS exposure and change in exposure | Measured from baseline through 5, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne F. Hovell, Study Chair — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States